CLINICAL TRIAL: NCT01056536
Title: Efficacy of a Brief Intervention and/or Distribution of Free Condoms During Pre-travel Consultation on Sexual Behaviour Abroad: a Randomized Controlled Trial
Brief Title: Brief Intervention and/or Distribution of Free Condoms for Travelers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Lausanne Hospitals (Other)
Responsible Party: Principal Investigator, Serge de Valliere, Consultant, University of Lausanne Hospitals
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MST
Record Dates: First submitted 2010-01-25; First posted 2010-01-26 (Estimated); Results first posted 2020-03-24 (Actual); Last update posted 2020-03-24 (Actual); Status verified 2020-03

CONDITIONS: Sexually Transmitted Infections
Keywords: Travel; casual sexual relationships; condoms; Structured intervention
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Structured intervention + free condoms (Experimental): The subjects will receive a structured intervention on STI's and will be offered free condoms
  Interventions: Behavioral: Structured intervention for the prevention of sexually transmitted infections (STI).; Device: Free condoms
- Free condoms (Active Comparator): Subjects will be offered free condoms at the end of the pre-travel consultation
  Interventions: Device: Free condoms
- No intervention (No Intervention): The topic of STI's will not be actively discussed during the pretravel consultation

INTERVENTIONS:
Behavioral: Structured intervention for the prevention of sexually transmitted infections (STI). — The structured intervention will include information about the number of travelers engaging in new sexual relationships, the different types of STI and their prevalence in different countries and population groups. The intervention will last approximately 5 minutes. At the end of the structured intervention the subjects will be offered free condoms.
  Arms: Structured intervention + free condoms
Device: Free condoms — Subjects will be proposed free condoms at the end of the pre-travel consultation.
  Arms: Free condoms; Structured intervention + free condoms

SUMMARY:
The objective of this study is to assess the impact of a structured intervention and/or free distribution of condoms during the pre-travel consultation on sexual risk behavior of young persons traveling alone.

DETAILED DESCRIPTION:
All persons aged 18 - 44 years planning to travel alone and attending the travel clinic of the Medical Outpatient Clinic in Lausanne will be asked to participate. The subjects will be randomized into three groups: 1. no intervention, 2. free condoms without further explanations, 3. a structured intervention of 5 minutes on STI risk reduction plus free condoms. The structured interventions will include information about the number of travelers engaging in new sexual relationships, the different types of STI and their prevalence in different countries and population groups. The subjects will complete a pre-travel questionnaire prior to the medical consultation. A post-travel questionnaire will be sent to them 10 days after their trip. The questionnaires will include questions on demographic characteristics, sexual habits, alcohol/tobacco/marijuana consumption and sexual relationships during the trip.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 - 44 years
* Travelling without the regular partner

Exclusion Criteria:

* Refusal of patient to participate

Ages: 18 Years to 44 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1681 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Travel Clinic, Medical Outpatient Department, University of Lausanne, Lausanne, Canton of Vaud, Switzerland

REFERENCES:
- [Derived] Senn N, de Valliere S, Berdoz D, Genton B. Motivational brief intervention for the prevention of sexually transmitted infections in travelers: a randomized controlled trial. BMC Infect Dis. 2011 Nov 1;11:300. doi: 10.1186/1471-2334-11-300. PMID 22044609

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were recruited between January 2006 and December 2008.The study was proposed by the administrative staff in the waiting room of the travel clinic.
Pre-assignment Details: The study was proposed to 5148 eligible travelers. 1681 travelers accepted to complete the pre-travel questionnaire. 1115 travelers completed the post-travel questionnaire.
Groups:
- Structured Intervention + Free Condoms: The subjects will receive a structured intervention on STI's and will be offered free condoms
  Structured intervention for the prevention of sexually transmitted infections (STI): The structured intervention will include information about the number of travelers engaging in new sexual relationships, the different types of STI and their prevalence in different countries and population groups. The intervention will last approximately 5 minutes. At the end of the structured intervention the subjects will be offered free condoms.
- Free Condoms: Subjects will be offered free condoms at the end of the pre-travel consultation
  Structured intervention for the prevention of sexually transmitted infections (STI): The structured intervention will include information about the number of travelers engaging in new sexual relationships, the different types of STI and their prevalence in different countries and population groups. The intervention will last approximately 5 minutes. At the end of the structured intervention the subjects will be offered free condoms.
Period: Overall Study
Arm/Group | Structured Intervention + Free Condoms | Free Condoms | No Intervention
Started | 596 | 356 | 729
Completed | 394 | 240 | 481
Not Completed | 202 | 116 | 248
Not completed — Lost to Follow-up | 202 | 116 | 248

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Structured Intervention + Free Condoms | Free Condoms | No Intervention | Total
Number analyzed (Participants) | 394 | 240 | 481 | 1115
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 394 | 240 | 481 | 1115
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 210 | 113 | 262 | 585
  Male | 184 | 127 | 219 | 530
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Switzerland | 394 | 240 | 481 | 1115

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Had New Sexual Relationships
Time Frame: 10 days after returning from abroad
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Intervention + Free Condoms | Free Condoms | No Intervention
Number analyzed (Participants) | 394 | 240 | 481
Participants | 56 | 37 | 61

2. Secondary Outcome: Number of Subjects Who Used Condoms Inconsistently
Time Frame: 10 days after returning from abroad
Measure: Count of Participants; unit: Participants
Arm/Group | Structured Intervention + Free Condoms | Free Condoms | No Intervention
Number analyzed (Participants) | 394 | 240 | 481
Participants | 11 | 10 | 14

ADVERSE EVENTS:
Arm/Group | Structured Intervention + Free Condoms | Free Condoms | No Intervention
Serious Adverse Events (participants affected / at risk) | 0/394 | 0/240 | 0/481
Other Adverse Events (participants affected / at risk) | 0/394 | 0/240 | 0/481

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No